## STATISTICAL ANALYSIS PLAN

STUDY TITLE: BOOSTER EFFECTS WITH AUTOIMMUNE TREATMENTS IN PARTICIPANTS WITH POOR RESPONSE TO INITIAL COVID-19 VACCINE

PROTOCOL NUMBER: ACV01

SHORT TITLE: COVID-19 BOOSTER VACCINE IN AUTOIMMUNE DISEASE

NON-RESPONDERS

NCT#: NCT05000216

CLIENT: The National Institute of Allergy and Infectious Diseases (NIAID)

REGULATORY

AGENCY IND# 27528

IDENTIFIER
NUMBER(S):

PREPARED BY:



This document is confidential and proprietary to NIAID. This study is being conducted in compliance with good clinical practice, including the archiving of essential documents. Acceptance of this document constitutes agreement by the recipient that no unpublished information contained herein will be reproduced, published, or otherwise disclosed without the prior written approval of NIAID, except that this document may be disclosed to appropriate Institutional Review Boards under the condition that they keep the information confidential.

# ACKNOWLEDGEMENT AND SIGNATURE SHEET

| Approved: | Approved: |
|---------------------------|---------------------------------|
| Principal Biostatistician | Principal Statistical Scientist |
| Signature and Date | Signature and Date |

| Approved: | Approved: |
|--------------------|--------------------|
| Medical Monitor | Medical Monitor |
| Signature and Date | Signature and Date |

| Approved: | Approved: |
|-----------------------|-----------------------|
| Judith James, MD, PhD | Meggan Mackay, MD, MS |
| Protocol Co-Chair | Protocol Co-Chair |
| Signature and Date | Signature and Date |


| Approved: | Approved: |
|--------------------------|------------------------|
| Dinesh Khanna, MBBS, MSC | Amit Bar-Or, MD, FRCPC |
| Protocol Co-Chair | Protocol Co-Chair |
| Signature and Date | Signature and Date |

| Approved: | Approved: |
|----------------------|--------------------|
| Virginia Pascual, MD | Stacy Ardoin, MD |
| Protocol Co-Chair | Protocol Co-Chair |
| Signature and Date | Signature and Date |

| Approved: | Approved: |
|---------------------------|--------------------|
| Natasha Mckerran Ruth, MD | Tracey Wright, MD |
| Protocol Co-Chair | Protocol Co-Chair |
| Signature and Date | Signature and Date |

# **VERSION HISTORY**

| SAP Version | Version Date | Change(s) | Rationale |
|-------------|--------------|---------------|-----------|
| 0.1 | 02Mar2022 | Initial Draft | |
| 1.0 | 16Mar2022 | Final Draft | |

## **TABLE OF CONTENTS**

| 1. | LIST OF ABBREVIATIONS | 8 |
|--------|------------------------------------------------|----|
| 2. | PURPOSE OF THE ANALYSES | 10 |
| 3. | PROTOCOL SUMMARY | 11 |
| 4. | GENERAL ANALYSIS AND REPORTING CONVENTIONS | 30 |
| 5. | ANALYSIS SAMPLES | 31 |
| 6. | STUDY SUBJECTS | 32 |
| 6.1. | Disposition of Subjects | 32 |
| 6.2. | Demographic and Other Baseline Characteristics | 32 |
| 6.3. | Prior and Concomitant Medications | 33 |
| 6.4. | Medical History | 33 |
| 7. | STUDY OPERATIONS | 34 |
| 7.1. | Protocol Deviations | 34 |
| 7.2. | Randomization and Allocation | 34 |
| 7.2.1. | Adult Stage 1 | 34 |
| 7.2.2. | Adult Stage 2 | 34 |
| 7.2.3. | Pediatric Population | 35 |
| 7.3. | Measures of Treatment Compliance | 35 |
| 8. | ENDPOINT EVALUATION | 36 |
| 8.1. | Overview of Efficacy Analysis Methods | 36 |
| 8.1.1. | Multicenter Studies | 36 |
| 8.1.2. | Assessment Time Windows | 36 |
| 8.1.3. | Timing of Analyses | 36 |
| 8.1.4. | Multiple Comparisons/Multiplicity | 36 |
| 8.2. | Primary Endpoint | 36 |
| 8.2.1. | Computation of the Primary Endpoint | 36 |
| 8.2.2. | Primary Analysis of the Primary Endpoint | 37 |
| 8.2.3. | Sensitivity Analyses of the Primary Analysis | 37 |
| 8.2.4. | Secondary Analyses of the Primary Endpoint | 37 |
| 8.3. | Secondary Endpoints | 38 |
| 8.3.1. | Seroconversion at Week 4 | 38 |

# The National Institute of Allergy and Infectious Diseases (NIAID) Statistical Analysis Plan - Protocol ACV01

| 8.3.2. | Fold Increase in anti-COVID-19 Antibody Levels at Week 4 | 39 |
|---|---|---|
| 8.3.3. | Longitudinal Changes in anti-COVID-19 Antibody Responses | 39 |
| 8.3.4. | Longitudinal Changes in Neutralization and Pseudo Neutralization Assays | 39 |
| 8.3.5. | Changes in Diseases Activity using CGI-C | 40 |
| 8.3.6. | Changes in Diseases Activity using PGA | 40 |
| 8.3.7. | Changes in Disease Activity as Measured by Disease-Specific Assessments | 40 |
| 8.3.8. | Changes in Patient-reported Outcomes | 41 |
| 8.4. | Other Endpoints | 42 |
| 8.5. | Examination of Subgroups | 42 |
| 9. | SAFETY EVALUATION | 43 |
| 9.1. | Overview of Safety Analysis Methods | 43 |
| 9.2. | Adverse Events | 43 |
| 9.2.1. | Solicited Adverse Events | 45 |
| 9.3. | Deaths, Serious Adverse Events, and Other Significant Adverse Events | 45 |
| 9.4. | Clinical Laboratory Evaluation | 46 |
| 9.5. | Vital Signs, Physical Findings, and Other Observations Related to Safety | 46 |
| 9.5.1. | Vital Signs | 46 |
| 9.5.2. | Physical Examinations | 46 |
| 9.5.3. | Other Safety Measures | 46 |
| 10. | OTHER ANALYSES | 47 |
| 11. | INTERIM ANALYSES AND DATA MONITORING | 48 |
| 12. | CHANGES TO THE ANALYSES PLANNED IN THE PROTOCOL | 49 |
| 13. | REFERENCES | 50 |
| 14. | APPENDIX | 51 |
| 14.1. | Study Flow Chart | 51 |
| 14.2. | Schedule of Events | 54 |
| 15 | ATT A CHMENTS | 55 |

## The National Institute of Allergy and Infectious Diseases (NIAID) Statistical Analysis Plan - Protocol ACV01

## LIST OF TABLES

| Table 1: | List of Abbreviations | .8 |
|----------|-----------------------|----|
|----------|-----------------------|----|

## 1. LIST OF ABBREVIATIONS

**Table 1: List of Abbreviations** 

| Abbreviation | Term |
|--------------|------------------------------------------------------------|
| ACE | Autoimmunity Centers of Excellence |
| AE | Adverse event |
| CRF | Case report forms |
| CSR | Clinical Study Report |
| CV | Coefficient of variation |
| DAIT | Division of Allergy, Immunology, and Transplantation |
| DAS | Disease Activity Score |
| DAS28-CRP | Disease Activity Score 28 using C-reactive protein |
| DSMB | Data and Safety Monitoring Board |
| EDSS | Expanded Disability Status Scale |
| H-SLEDAI | Hybrid Systemic Lupus Erythematosus Disease Activity Index |
| IS | Immunosuppressive medications |
| JADAS | Juvenile Arthritis Disease Activity Score |
| JDM | juvenile dermatomyositis |
| ЛА | juvenile idiopathic arthritis |
| LLOD | Lower Limit of Detection |
| MAAE | medically attended adverse event |
| MCAR | Missing-completely-at-random |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMF | Mycophenolate mofetil |
| MPA | Mycophenolic acid |
| MS | Multiple sclerosis |
| MTX | Methotrexate |
| NCI | National Cancer Institute |
| NIAID | The National Institute of Allergy and Infectious Diseases |
| NIH | National Institutes of Health |
| NOCMC | New onset chronic medical condition |
| PASI | Psoriasis Area and Severity Index |


# The National Institute of Allergy and Infectious Diseases (NIAID) Statistical Analysis Plan - Protocol ACV01

| PDAI | Pemphigus Disease Area Index |
|---|---|
| PedsQL | Pediatric Quality of Life Inventory™ |
| PGI-C | Patient Global Impression of Change |
| PtGA | Patient's Global Assessment |
| PGA | Physician Global Assessment |
| POMS | Pediatric-onset multiple sclerosis |
| PROMIS | Participant-Reported Outcomes Measurement Information System |
| PT | Preferred term |
| RA | Rheumatoid arthritis |
| RBD | Receptor binding domain |
| SACCC | Statistical and Clinical Coordinating Center |
| SAE | serious adverse event |
| SAP | Statistical analysis plan |
| SARS-COV-2 | Severe Acute Respiratory Syndrome Coronavirus-2 |
| SD | Standard deviation |
| SARS-COV-2 | Severe Acute Respiratory Syndrome Coronavirus-2 |
| SELENA-<br>SLEDAI | Safety of Estrogens in Lupus Erythematosus: National Assessment– Systemic<br>Lupus Erythematosus Disease Activity Index |
| SLE | Systemic lupus erythematosus |
| SOC | System organ class |
| SSc | Systemic sclerosis |
| VRC | Vaccine Research Center |
| WHO | World Health Organization |

#### 2. PURPOSE OF THE ANALYSES

The purpose of this statistical analysis plan (SAP) is to describe the planned analyses and data displays to be included in the Clinical Study Report (CSR) for Protocol ACV01. This document provides details on study populations, how the variables will be derived, how missing data will be handled and details on statistical methods to be used to analyze the safety and efficacy data.

The SAP is based on ICH guidelines E3 and E9 (Statistical Principles for Clinical Trials).

The document will be updated over time to reflect the requirements of the adaptive study design, protocol amendments and any regulatory requests. However, the final SAP must be finalized, approved by the Client, and placed on file before database is locked. If differences occur between analyses described in the SAP and the current protocol, those found in this SAP will assume primacy. Deviations from the final approved plan will be noted in the clinical study report.

Document Control No.: TMP-SA-008-01 Template Effective Date: 23 Mar 2021

Version: 1.0

## 3. PROTOCOL SUMMARY

Version 1.0 of the protocol was finalized July 9, 2021; the protocol is currently under Version 3.0 which includes several of the planned adaptive elements to ACV01, and is summarized below.

| Title | Booster effects with autoimmune treatments in patients with poor response to initial COVID-<br>19 vaccine |
|---|---|
| Short Title | COVID-19 BOOSTER VACCINE IN AUTOIMMUNE DISEASE NON-<br>RESPONDERS |
| Clinical Phase | п |
| Number of Sites | Adult population: 15 – 20 sites in the United States (US) that are active National Institute of Allergy and Infectious Diseases (NIAID) Autoimmunity Centers of Excellence (ACE) or active subaward recipients of the NIAID ACE Network Pediatric population: 15 – 20 sites in the US. |
| IND Sponsor/Number | The National Institute of Allergy and Infectious Diseases (NIAID) / IND #27528 |
| Study Objectives | Hypotheses We hypothesize that adult and pediatric participants with autoimmune diseases requiring immunosuppressive (IS) medications who have had a sub-optimal response to an initial COVID-19 vaccine regimen may demonstrate enhanced immune response after receiving an additional homologous dose of an mRNA or vector-based vaccine. We hypothesize that adult and pediatric participants with transient cessation of mycophenolate mofetil (MMF)/ mycophenolic acid (MPA) or methotrexate (MTX) before and after vaccination will have an enhanced immune response. We further hypothesize that adult participants with autoimmune diseases requiring IS medications who continue to have a sub-optimal response after an initial COVID-19 vaccine regimen plus an additional homologous vaccine dose may demonstrate enhanced immune response after receiving an additional dose of an alternative COVID-19 vaccine. Primary Objective The primary objective is to determine the proportions of adult and pediatric participants who have a protective antibody response at 4 weeks after an additional homologous dose of a COVID-19 vaccine using the NIAID Vaccine Research Center (NIAID-VRC) MSD 3 plex (Wu-1 full-length spike, RBD, and N proteins) assay within arms defined by the initial COVID-19 vaccine regimen received, IS regimens, and treatment plans to either withhold or continue medications around the time of vaccination. Secondary Objectives Stage 1 Secondary Objectives (adult & pediatric): |

- To determine the incidence of seroconversion following an additional homologous COVID-19 vaccine dose in the subgroup of participants that are anti-COVID-19 antibody negative at Baseline.
- To determine the incidence of adverse events (AEs), including medically attended
  adverse events (MAAEs), new onset chronic medical conditions (NOCMCs), and
  serious adverse events (SAEs) following an additional homologous COVID-19
  vaccine dose.
- To assess whether responses to an additional homologous COVID-19 vaccine dose differ with temporary cessation of IS medications around the time of vaccine.
- To assess whether responses to an additional homologous COVID-19 vaccine dose differ by type of vaccine administered.
- To assess whether responses to an additional homologous COVID-19 vaccine dose differ by type of cohort-defining IS medications and by disease type.
- To assess whether response to an additional homologous COVID-19 vaccine dose is associated with corticosteroid dose at the time of vaccination.
- To assess whether response to an additional homologous COVID-19 vaccine dose is associated with clinical parameters including disease activity, co-morbid illness, age, and sex.
- To determine whether disease activity is increased following an additional homologous COVID-19 vaccine dose, and if so, whether Baseline or induced immunologic variables are associated with increased disease activity and/or vaccination response.

#### Stage 2 Secondary Objectives (adult):

- To determine the proportions of participants with a negative serologic or sub-optimal response to an additional homologous COVID-19 vaccine dose who develop a protective antibody response after receiving a subsequent alternative vaccine dose, evaluated using the NIAID-VRC MSD 3 plex (Wu-1 full-length spike, RBD, and N proteins) assay.
- To determine the incidence of seroconversion following a subsequent alternative vaccine dose in the subgroup of participants that are anti-COVID-19 antibody negative following an additional homologous COVID-19 vaccine dose.
- To determine the incidence of AEs, including MAAEs, NOCMCs, and SAEs following a subsequent alternative COVID-19 vaccine dose.
- To assess whether responses to a subsequent alternative COVID-19 vaccine dose differ by type of vaccine administered.
- To assess whether responses to a subsequent alternative COVID-19 vaccine dose differ by type of cohort-defining IS medications and by disease type.


- To assess whether response to a subsequent alternative COVID-19 vaccine dose is associated with corticosteroid dose at the time of vaccination.
- To assess whether response to a subsequent alternative COVID-19 vaccine dose is associated with clinical parameters including disease activity, co-morbid illness, age, and sex
- To determine whether disease activity is increased following a subsequent alternative COVID-19 vaccine dose, and if so, whether immunologic variables are associated with increased disease activity and/or vaccination response.

#### **Exploratory Objectives:**

- To evaluate whether Baseline CD19 positive B cell numbers associate with response to an additional study COVID-19 vaccine dose in the cohort that have received B cell depletion therapy.
- To evaluate the association between immune response and levels of SARS-CoV-2 antibodies at Baseline.
- To evaluate the levels of Baseline interferon signal or interferon gamma-inducible protein 10 (IP-10) serum levels that associate with an effective vaccine response.
- To evaluate the levels of Baseline inflammatory signals that associate with an effective vaccine immune response.
- To evaluate the association between immune response to an additional study COVID-19 vaccine dose and cellular and mechanistic endpoints.

#### Study Design

This is a randomized, multi-site, adaptive, open-label clinical trial comparing the immune response to different additional doses of COVID-19 vaccine in participants with autoimmune disease requiring IS medications. All study participants will have negative serologic or suboptimal responses (defined as a Roche Elecsys® Anti-SARS-CoV-2 S result ≤200 U/mL) to initial COVID-19 vaccine regimen with Moderna COVID-19 Vaccine, Pfizer-BioNTech COVID-19 Vaccine, or Janssen COVID-19 Vaccine.

#### **Adult Population:**

#### Adult Stage 1:

Stage 1 of this trial will enroll up to a maximum of 900 adult study participants (up to 60 participants per arm). The trial initially focused on adults with at least 1 of 5 autoimmune diseases: systemic lupus erythematosus (SLE), rheumatoid arthritis (RA), multiple sclerosis (MS), systemic sclerosis (SSc), and pemphigus.

Participants will be assigned to one of 3 cohorts based on their IS regimens:

- Cohort A: Receipt of MMF or MPA
- Cohort B: Receipt of MTX
- Cohort C: Receipt of any B cell depletion therapy within the past 18 months.

*Treatment Arms:* Participants in Cohorts A, B, and C will be assigned to receive an additional dose of the same vaccine as their original vaccine series.

Participants in Cohorts A and B will be randomized into two IS medication treatment plans as follows

- Participants continue to take their cohort-defining IS medications without alterations in schedule and dosing.
- Participants withhold their cohort-defining IS medications before and after the additional homologous vaccine dose per protocol instructions.


Schedule of Events: Visits to assess endpoints will occur at Baseline (Week 0), Week  $4 \pm 1$  week, Week  $12 \pm 2$  weeks, Week  $24 \pm 2$  weeks, Week  $36 \pm 2$  weeks, and Week  $48 \pm 2$  weeks. A participant will be enrolled in the study for a maximum of approximately 13 months.

#### Adult Stage 2:

Stage 2 of this trial will include up to a maximum of 540 adult study participants (up to 60 per arm). Participants will be eligible to receive a dose of an alternative COVID-19 vaccine. Participants may have received their additional homologous vaccine dose as a Stage 1 study participant and then enter into Stage 2 ("rollover participant"), or they may have received their additional homologous dose prior to enrollment in the study ("newly recruited participant").

Participants will be allocated to 1 of 3 cohorts based on their IS regimens:

- Cohort D: Receipt of MMF or MPA
- Cohort E: Receipt of MTX
- Cohort F: Receipt of any B cell depletion therapy within the past 18 months.

Treatment Arms: Participants in Cohorts D, E, and F will receive a dose of an alternative COVID-19 vaccine compared to their previous COVID-19 vaccine doses. Participants who previously received 3 total doses of an mRNA vaccine (Moderna COVID-19 Vaccine OR Pfizer-BioNTech COVID-19 Vaccine) will receive their choice of either the Janssen vector-based COVID 19 vaccine or the other mRNA COVID-19 vaccine, and participants who previously received 2 doses of the Janssen vector-based COVID-19 vaccine will receive the Moderna COVID-19 Vaccine.

Participants in Cohorts D and E will withhold their cohort-defining IS medications before and after the alternative vaccine dose per protocol instructions. Participants in Cohort F who are taking MMF, MPA, or MTX in addition to B cell depletion therapies (BCDTs) will withhold these medications before and after the alternative vaccine dose per protocol instructions. Schedule of Events: Visits to assess endpoints will occur at Baseline (Week 0), Week  $4 \pm 1$  week, Week  $12 \pm 2$  weeks, Week  $24 \pm 2$  weeks, Week  $36 \pm 2$  weeks, and Week  $48 \pm 2$  weeks. A participant who enters Stage 2 after a serologic negative or sub-optimal response to their Stage 1 vaccine dose may be on study for up to a maximum of 26 months. A participant who is newly recruited to the study for entry into Stage 2 may be on study for up to a maximum of 13 months.

#### **Pediatric Population:**

The pediatric portion of this trial will enroll up to a maximum of 900 participants (5-17 years of age) with a Roche Elecsys® Anti-SARS-CoV-2 S result ≤200 U/mL after receiving an initial COVID-19 vaccine regimen (up to 60 participants per arm). Vaccines will be included in this protocol as they receive EUA or approval by FDA for a given age group. Pediatric participants will have 1 of 4 autoimmune diseases: pediatric SLE, juvenile idiopathic arthritis (JIA), juvenile dermatomyositis (JDM), or pediatric-onset multiple sclerosis (POMS). Participants will be assigned to one of 3 cohorts based on their IS regimens:

- Cohort A: Receipt of MMF or MPA
- Cohort B: Receipt of MTX
- Cohort C: Receipt of any B cell depletion therapy within the past 18 months.

*Treatment Arms:* Participants in Cohorts A, B, and C will be assigned to receive an additional dose of the same vaccine as their original vaccine series.

Participants in Cohorts A and B will be randomized into two IS medication treatment plans as follows):

 Participants continue to take their cohort-defining IS medications without alterations in schedule and dosing.

| | Participants withhold their cohort-defining IS medications before and after the |
|---|---|
| | additional homologous vaccine dose per protocol instructions. |
| | Schedule of Events: Visits to assess endpoints will occur at Baseline (Week 0), Week 4 ± 1 week, Week 12 ± 2 weeks, Week 24 ± 2 weeks, Week 36 ± 2 weeks, and Week 48 ± 2 weeks. A participant will be enrolled in the study for a maximum of approximately 13 months. Adaptive Design: An adaptive design will be employed such that cohorts and arms defined by additional vaccine doses and IS treatment plans may be added or modified based on emerging data from existing and new FDA Emergency Use Authorization (EUA) or approvals of COVID-19 vaccines: |
| | <ul> <li>New cohorts may be defined based on changes in the medication groups if it<br/>becomes obvious that certain medications are highly associated with sub-optimal<br/>serologic response to initial COVID-19 vaccine regimen.</li> </ul> |
| | <ul> <li>Cohorts may limit or expand the autoimmune diseases that are eligible to be<br/>included in the clinical trial, and may include expansion cohorts of underrepresented<br/>diseases.</li> </ul> |
| | New cohorts may include participants whose antibody response falls to sub-optimal levels over time. |
| | Based upon timing of the FDA EUA authorization for children of each of the COVID-19 vaccines used in this trial, the age range of the inclusion criteria may be expanded. |
| | Allocation or randomization to treatment with new vaccines designed for COVID variants or with a protein-based vaccine may be incorporated into the design when the products become available. |
| | Identification of additional strategies to enhance vaccine responsiveness in autoimmune diseases, including a temporary switch of immunomodulatory medications. |
| Primary Endpoint | The primary endpoint in the adult and pediatric populations of a protective antibody response at Week 4 will be assessed by the NIAID-VRC MSD 3 plex (Wu-1 full-length spike, RBD, and N proteins) assay. |
| Secondary and<br>Exploratory<br>Endpoints | Secondary Endpoints Secondary endpoints related to antibody response will primarily be assessed by the NIAID-VRC MSD 3 plex (Wu-1 full-length spike, RBD, and N proteins) assay; where applicable, they will also be assessed by the Roche Elecsys® Anti-SARS-CoV-2 S electrochemiluminescence immunoassay. |
| | The secondary endpoints are applicable to both the adult and pediatric populations. • Seroconversion at Week 4 following additional doses of COVID-19 vaccine in the subgroup of participants that are anti-COVID-19 antibody negative at Week 0. |


- Fold increase in anti-COVID-19 antibody levels at Week 4 following an additional dose of COVID-19 vaccine in the subgroup of participants who are anti-COVID-19 antibody positive at Week 0.
- Longitudinal changes in anti-COVID-19 antibody responses from Week 0 to Weeks 4, 12, 24, 36, and 48.
- Longitudinal changes in neutralization and pseudo neutralization assays from Week
   to Weeks 4, 12, 24, 36, and 48.
- Changes in disease activity after receipt of additional doses of COVID-19 vaccine as measured by the Clinical Global Impression of Change (CGI-C).
- Changes in disease activity after receipt of additional doses of COVID-19 vaccine as measured by the Physician Global Assessment (PGA).
- Changes in disease activity after receipt of additional doses of COVID-19 vaccine as measured by the following disease-specific assessments:
  - o Adult population disease assessments:
    - Hybrid Systemic Lupus Erythematosus Disease Activity Index (H-SLEDAI) and Thanou modified Safety of Estrogens in Lupus Erythematosus: National Assessment

       – Systemic Lupus
       Erythematosus Disease Activity Index (SELENA-SLEDAI) Flare
       Index for SLE
    - Disease Activity Score 28 using C-reactive protein (DAS28-CRP) for RA
    - Flare assessment for SSc (including patient reported flare assessment)
    - o Pemphigus Disease Area Index (PDAI) for pemphigus
    - Physician-assessed relapse for MS
  - o Pediatric population disease assessments:
    - о ЛА:
      - JADAS10 for polyarthritis, enthesitis related to JIA, oligoarthritis, and psoriatic arthritis
      - Psoriasis Area and Severity Index (PASI) for psoriatic arthritis
    - SLEDAI-2K and Childhood-onset SLE Criteria for Global Flare
       [1] for pediatric SLE
    - Childhood Myositis Assessment Scale (CMAS) and JDM Disease Activity Score (DAS) for JDM
    - Physician-assessed relapse for MS for POMS

- Changes in patient-reported outcomes as measured by:
  - Participant-Reported Outcomes Measurement Information System (PROMIS) 29 (adults only)
  - o Pediatric Quality of Life Inventory™ (PedsQL) (pediatrics only)
  - o Patient Global Assessment (PtGA)
  - o Patient Global Impression of Change (PGI-C)
- The proportion of participants who experience the following safety events:
  - Any Grade 1 or higher AEs related to the additional doses of COVID-19 vaccine
  - o Any SAEs, MAAEs, NOCMCs
  - o Any SARS-CoV-2 infection

#### **Exploratory Endpoints**

- Changes in autoantibody levels after COVID-19 vaccination between Week 0, and Weeks 4, 12, 24, 36, and 48.
- Assessments of cellular and mechanistic response, including
  - o Immune cell population profiling over time
  - o Antigen-specific T cell responses
  - o Antigen-specific memory B cell responses
  - o Total IgG responses
  - o B cell and T cell repertoire
  - o Changes in gene expression profile modules
  - o Plasma levels of soluble mediators

#### **Accrual Objective**

#### **Adult Population:**

In Stage 1, 15 arms are planned within cohorts defined by categories of IS medications such that a maximum of 900 participants are to be randomized/allocated. In Adult Stage 2, 9 arms are planned to evaluate the immune response to a subsequent alternative COVID-19 vaccine dose such that a maximum of 540 participants (either rollover or newly recruited) are to be allocated.

#### **Pediatric Population:**

A total of 15 arms are planned within cohorts defined by categories of IS medications such that a maximum of 900 participants are to be randomized/allocated (up to 300 participants for each vaccine to receive FDA EUA in pediatric participants).

In all populations and stages, 40 participants with a Roche Elecsys® Anti-SARS-CoV-2 S result ≤50 U/mL will be targeted for each arm, with a total of 60 participants with a Roche Elecsys® Anti-SARS-CoV-2 S result ≤200 U/mL randomized or allocated to each arm. In each arm, the number of participants with Roche Elecsys® Anti-SARS-CoV-2 S results ≤50 U/mL will be capped at 40 participants, and the number of participants with Roche Elecsys® Anti-SARS-CoV-2 S results >50 U/mL and ≤200 U/mL will be capped at 40 participants.

| Study Duration | Study duration for Adult Stage 1, Adult Stage 2 newly recruited, or pediatric participant: 13 months Study duration for Adult 2 participant rolling over from Stage 1: maximum of 26 months |
|---|---|
| Treatment<br>Description | All participants will receive one dose of the following: mRNA COVID-19 vaccine: Moderna OR mRNA COVID-19 vaccine: Pfizer-BioNTech OR vector-based COVID-19 vaccine: Janssen |
| Inclusion/Exclusion<br>Criteria – Adult Stage<br>1 | <ol> <li>Inclusion Criteria: Individuals who meet all of the following criteria are eligible for randomization/allocation as study participants in Adult Stage 1: </li> <li>Individuals 18 years of age or older that meet classification criteria for SLE, SSc, RA, MS, or pemphigus.</li> <li>Participants must meet the 2019 ACR/EULAR[2] or 2012 SLICC classification criteria for SLE [3], the 2010 ACR/EULAR classification criteria for RA [4], the 2013 EULAR/ACR classification criteria for SSc [5], the 2017 McDonald [6] criteria for MS, and the international consensus criteria for pemphigus [7].</li></ol> |
| | b. If enrolling in the B cell depleting therapy cohort, the participant must have<br>received an anti-CD20 or an anti-CD19 B cell depleting therapy in the past 18<br>months. |


- 7. No changes in background IS medications, including MMF/MPA or MTX, in the 8 weeks prior to Screening, excluding the following:
  - a. HCQ,
  - b. Intraarticular steroids,
  - c. The addition of prednisone at ≤10mg per day or prednisone at any dose when given for ≤3 days, and
  - d. Corticosteroid bursts for non-autoimmune disease-related conditions, such as asthma or COPD, are permitted.

#### **Exclusion Criteria:**

Individuals who meet any of these criteria are not eligible for randomization/allocation as study participants in Adult Stage 1:

- Inability or unwillingness of a participant to give written informed consent or comply with study protocol.
- 2. History of severe allergic reaction to the initial COVID-19 vaccine regimen, to any component of any of the COVID-19 vaccines, or to polyethylene glycol (PEG).
- 3. New diagnosis of malignancy that will require chemotherapy or immunotherapy, or ongoing treatment for a malignancy with chemotherapy or immunotherapy.
- 4. Active disease (per the Investigator's decision) resulting in inability to hold the IS therapy in the MMF/MPA or MTX arms of the study.
  - a. The potential impact of temporarily holding medication for participants with a recent mild disease flare within 4 weeks should be carefully considered.
- 5. Active disease during the Screening period resulting in:
  - a. An increase/addition of IS medications, or
  - b. A suggestion of MS relapse per the investigator
- 6. Recent or current SARS-CoV-2 infection defined as:
  - a. Documented SARS-CoV-2 infection in the past 30 days (from the day the participant is diagnosed by positive test to Screening).
  - b. Positive result on a molecular COVID-19 test at Screening.
- Receipt of a COVID-19 vaccine booster prior to Screening with the Moderna COVID-19 Vaccine, Pfizer-BioNTech COVID-19 Vaccine, or Janssen COVID-19 Vaccine.
- Inflammatory myocarditis/pericarditis following initial COVID-19 vaccine regimen.
- Participants with active, ongoing chronic infections, including participants with evidence of:
  - a. Human Immunodeficiency Virus (HIV)
  - b. Hepatitis B as indicated by surface antigen

| | c. Hepatitis C as indicated by anti-hepatitis C antibody positivity; if a participant is Hepatitis C antibody positive, they will be eligible to participate in the study if he/she is negative for viral load at Screening. Note: Participants are permitted to be on chronic prophylactic antimicrobial therapy. |
|---|---|
| | <ol> <li>Participants with common variable immunodeficiency disease, as well as any<br/>participants currently receiving immune globulin replacement therapy.</li> </ol> |
| | <ol> <li>Participants who received licensed or investigational monoclonal antibodies or<br/>plasma products directed against SARS-CoV-2 within 30 days of Screening.</li> </ol> |
| | 12. Participants who have received any live vaccines within 2 months of the anticipated study vaccine dose or who will have need of a live vaccine at any time during the study. |
| | 13. Currently pregnant or breastfeeding. |
| | 14. Participants who are planning a pregnancy during the course of the trial. |
| | 15. Hemoglobin (Hgb) <8.0 g/dL (80 g/L) |
| | 16. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study. |
| | 17. Other investigational chemical agent within 30 days or other investigational biologic agent within 8 weeks or 5 half-lives (whichever is longer) of Screening. |
| | <ol> <li>Concurrent treatment with cyclophosphamide, cladribine, alemtuzumab, or<br/>mitoxantrone.</li> </ol> |
| | <ol> <li>Participants currently on any type of dialysis, or who have received a solid organ<br/>transplant.</li> </ol> |
| | <ol> <li>Prisoners or participants who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness.</li> </ol> |
| | 21. Taking both MMF/MPA and MTX. |
| | <ol> <li>Receiving other investigational B cell depleting therapy as part of a clinical trial within 18 months of Screening, unless drug assignment is known and the participant received an anti-CD20 or CD19 drug.</li> </ol> |
| | <ol> <li>Participants with active systemic infections who have received systemic<br/>antimicrobials within the 14 days prior to Screening.</li> </ol> |
| Inclusion/Exclusion<br>Criteria – Adult Stage<br>2 Newly Recruited | Inclusion Criteria: Individuals who meet all of the following criteria are eligible for enrollment as participants in Stage 2: |


**Participants** 

Version Date: 2022-03-16 Version: 1.0

- Individuals 18 years of age or older that meet classification criteria [1-6] for SLE, SSc, RA, MS, or pemphigus If a participant has been diagnosed with more than one autoimmune disease, the participant will be assessed based on the disease that is selected for study entry.
- 2. Willing and able to sign informed consent.
- Documented full COVID-19 vaccination (CDC card or documentation in medical records).
- Received an additional homologous COVID-19 vaccine dose (documented by CDC card or in medical records) that was completed at least 4 weeks prior and no more than 48 weeks prior to the Stage 2 Screening visit.
- Negative or suboptimal serologic response to the additional homologous COVID-19
  vaccine in one of the qualifying regimens, defined as an Elecsys® Anti-SARS-CoV2 S (RBD) negative result or positive result of ≤200 U/mL within 4 weeks of the
  Stage 2 Baseline/Week 0 visit.

The regimens of COVID-19 vaccination that qualify are as follows:

- a. 3 full doses of the Pfizer-BioNTech COVID-19 Vaccine
- b. 3 full doses of the Moderna COVID-19 Vaccine
- c. 2 full doses of the Janssen COVID-19 Vaccine
- 6. Must be currently taking one of the following IS medications with or without additional disease-related medications: MMF (minimum of 1000 mg per day)/MPA (minimum of 720 mg per day), MTX (minimum of 7.5mg per week), or B cell depleting agents within the past 18 months (such as rituximab, ocrelizumab, or ofatumumab).
  - a. If taking MMF/MPA or MTX, the participant must have initiated therapy at least 8 weeks prior to allocation and be taking the same medications (regardless of dose) as at the time of the initial COVID-19 vaccine regimen. Note: Participants who withheld their IS medications around their initial vaccinations are eligible to participate.
  - b. If enrolling in the B cell depleting therapy cohort, the participant must have received an anti-CD20 or an anti-CD19 B cell depleting therapy in the past 18 months.
- 7. No changes in background IS medications, including MMF/MPA or MTX, in the 4 weeks prior to Stage 2 Screening, excluding the following:
  - a. HCQ,
  - b. Intraarticular steroids,
  - c. The addition of prednisone at ≤10mg per day or prednisone at any dose when given for ≤3 days, and

d. Corticosteroid bursts for non-autoimmune disease-related conditions, such as asthma or COPD, are permitted.

#### **Exclusion Criteria:**

Individuals who meet any of these criteria are not eligible for randomization/allocation as study participants in Stage 2:

- Inability or unwillingness of a participant to give written informed consent or comply with study protocol.
- 2. History of severe allergic reaction to any previous COVID-19 vaccines, to any component of any of the COVID-19 vaccines, or to PEG.
- 3. New diagnosis of malignancy that will require chemotherapy or immunotherapy, or ongoing treatment for a malignancy with chemotherapy or immunotherapy.
- 4. Active disease (per the Investigator's decision) resulting in inability to hold the IS therapy in the MMF/MPA or MTX arms of the study.
  - a. The potential impact of temporarily holding medication for participants with a recent mild disease flare within 4 weeks should be carefully considered.
- 5. Active disease during the Stage 2 Screening period resulting in:
  - a. An increase/addition of any IS medications, or
  - b. A suggestion of MS relapse per the investigator.
- 6. Recent or current SARS-CoV-2 infection defined as:
  - Documented SARS-CoV-2 infection in the past 30 days (from the day the participant is diagnosed by positive test to Stage 2 Screening).
  - b. Positive result on a molecular COVID-19 test at Stage 2 Screening.
- Receipt of an additional heterologous COVID-19 vaccine dose prior to Stage 2
   Screening, i.e., a participant cannot have received a mixture of mRNA vaccines or both mRNA and Janssen COVID-19 vaccines in any order or combination.
- 8. Inflammatory myocarditis/pericarditis following any COVID-19 vaccine doses.
- Participants with active, ongoing chronic infections including participants with evidence of:
  - a. HIV.
  - b. Hepatitis B as indicated by surface antigen.
  - c. Hepatitis C as indicated by anti-hepatitis C antibody positivity; if a participant is Hepatitis C antibody positive, they will be eligible to participate in the study if he/she is negative for viral load at Stage 2 Screening.

Note: Participants are permitted to be on chronic prophylactic antimicrobial therapy.

- 10. Participants with common variable immunodeficiency disease, as well as any participants currently receiving immune globulin replacement therapy.
- Participants who received licensed or investigational monoclonal antibodies or plasma products directed against SARS-CoV-2 within 30 days of Stage 2 Screening.
- 12. Participants who have received any live vaccines within 2 months of the anticipated study vaccine dose or who will have need of a live vaccine at any time during the study.
- 13. Currently pregnant or breastfeeding.
- 14. Female participants who are planning a pregnancy during the course of the trial.
- 15. Hemoglobin (Hgb) <8.0 g/dL (80 g/L)
- 16. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.
- 17. Other investigational chemical agent within 30 days or other investigational biologic agent within 8 weeks or 5 half-lives (whichever is longer) of Stage 2 Screening.
- Concurrent treatment with cyclophosphamide, cladribine, alemtuzumab, or mitoxantrone.
- Participants currently on any type of dialysis, or who have received a solid organ transplant.
- 20. Prisoners or participants who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness.
- 21. Taking both MMF/MPA and MTX.
- 22. Receiving other investigational B cell depleting therapy as part of a clinical trial within 18 months of Screening, unless drug assignment is known and the participant received an anti-CD20 or CD19 drug.
- 23. Participants with active systemic infections who have received systemic antimicrobials within the 14 days prior to Stage 2 Screening.

## Inclusion/Exclusion Criteria – Adult Stage 2 Rollover Participants

#### **Inclusion Criteria:**

Individuals who meet all of the following criteria are eligible to continue as participants in Stage 2:

Negative or suboptimal serologic response to the additional homologous COVID-19
vaccine in one of the qualifying regimens, defined as an Elecsys® Anti-SARS-CoV-

2 S (RBD) negative result or positive result of ≤200 U/mL within 4 weeks of the Stage 2 Baseline/Week 0 visit.

The regimens of COVID-19 vaccination that qualify are as follows:

- a. 3 full doses of the Pfizer-BioNTech COVID-19 Vaccine
- b. 3 full doses of the Moderna COVID-19 Vaccine
- c. 2 full doses of the Janssen COVID-19 Vaccine
- 6. Must be currently taking one of the following IS medications with or without additional disease-related medications: MMF (minimum of 1000 mg per day)/MPA (minimum of 720 mg per day), MTX (minimum of 7.5mg per week), or B cell depleting agents within the past 18 months (such as rituximab, ocrelizumab, ofatumumab).
  - a. If taking MMF/MPA or MTX, the participant must have initiated therapy at least 8 weeks prior to allocation and be taking the same medications (regardless of dose) as at the time of the initial COVID-19 vaccine regimen. Note: Participants who withheld their IS medications around their initial vaccinations are eligible to participate.
  - b. If enrolling in the B cell depleting therapy cohort, the participant must have received an anti-CD20 or an anti-CD19 B cell depleting therapy in the past 18 months.
- 7. No changes in background IS medications, including MMF/MPA or MTX, in the 4 weeks prior to Stage 2 Baseline/Week 0 visit, excluding the following:
  - a. HCQ,
  - b. Intraarticular steroids,
  - c. The addition of prednisone at ≤10mg per day or prednisone at any dose when given for ≤3 days, and
  - d. Corticosteroid bursts for non-autoimmune disease-related conditions, such as asthma or COPD, are permitted.

#### **Exclusion Criteria:**

Individuals who meet any of these criteria are not eligible to continue as participants in Stage 2:

- 2. History of severe allergic reaction to any previous COVID-19 vaccines, to any component of any of the COVID-19 vaccines, or to PEG.
- 3. New diagnosis of malignancy that will require chemotherapy or immunotherapy, or ongoing treatment for a malignancy with chemotherapy or immunotherapy.
- 4. Active disease (per the Investigator's decision) resulting in inability to hold the IS therapy in the MMF/MPA or MTX arms of the study.

a. The potential impact of temporarily holding medication for participants with a recent mild disease flare within 4 weeks should be carefully considered. 5. Active disease during the Stage 2 Screening period resulting in: a. An increase/addition of any IS medications, or b. A suggestion of MS relapse per the investigator. 6. Recent or current SARS-CoV-2 infection defined as: a. Documented SARS-CoV-2 infection in the past 30 days (from the day the participant is diagnosed by positive test to Stage 2 Screening). b. Positive result on a molecular COVID-19 test at Stage 2 Screening or Stage 2 Baseline/Week 0. 8. Inflammatory myocarditis/pericarditis following any COVID-19 vaccine doses. 11. Participants who received licensed or investigational monoclonal antibodies or plasma products directed against SARS-CoV-2 within 30 days of Stage 2 Screening. 13. Currently pregnant or breastfeeding. 14. Female participants who are planning a pregnancy during the course of the trial. 15. Hemoglobin (Hgb) < 8.0 g/dL (80 g/L) 16. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study. 17. Other investigational chemical agent within 30 days or other investigational biologic agent within 8 weeks or 5 half-lives (whichever is longer) of Stage 2 Screening. 18. Concurrent treatment with cyclophosphamide, cladribine, alemtuzumab, or mitoxantrone. 19. Participants currently on any type of dialysis, or who have received a solid organ transplant. 20. Prisoners or participants who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness. 23. Participants with active systemic infections who have received systemic antimicrobials within the 14 days prior to Stage 2 Baseline/Week 0. Inclusion Criteria: Inclusion/Exclusion Criteria – Pediatric Individuals who meet all of the following criteria are eligible for enrollment **Participants** randomization/allocation as participants in the pediatric portion of the study:


- Individuals 5-17 years of age that meet classification criteria for SLE, JIA, POMS, or JDM. Note: Juvenile idiopathic arthritis includes the following conditions: polyarticular JIA (both RF + and -), oligoarticular persistent and oligoarticular extended JIA, psoriatic arthritis, and enthesitis related JIA.
  - a. Participants must meet the 2017 EULAR/ACR classification criteria for adult and juvenile idiopathic inflammatory myopathies and their major subgroups [8], the International League of Associations for Rheumatology (ILAR) classification for JIA [4], the 2017 McDonald [6] criteria for MS, or the Bohan and Peter criteria or the 2017 EULAR/ACR classification criteria for JDM.
  - b. If a participant has been diagnosed with more than one autoimmune disease, the participant will be assessed based on the disease that is selected for study entry.
- 2. Parents/guardians of pediatric participants must be willing and able to sign informed consent. Participants, ages 7-17, must be willing and able to sign assent.
- Documented full COVID-19 vaccination (CDC card or documentation in medical records) that was completed at least 4 weeks prior and no more than 52 weeks prior to the Screening visit.
- Negative or suboptimal serologic response to initial COVID-19 vaccine regimen, defined as an Elecsys® Anti-SARS-CoV-2 S result ≤200 U/mL at Screening visit.
  - a. Initial COVID-19 vaccine regimen is defined as:
    - i. 2 doses (as appropriate to age) of the Pfizer-BioNTech COVID-19 Vaccine

The following vaccines have yet to receive EUA in pediatric populations. If EUA occurs for younger ages, the participants receiving age-appropriate regimens of the following COVID-19 vaccines may be enrolled into the study:

- ii. Moderna COVID-19 Vaccine
- iii. Janssen COVID-19 Vaccine
- 5. Must be currently taking one of the following IS medications with or without additional disease-related medications: MMF (minimum of 250 mg per day)/MPA (minimum of 360 mg per day), MTX (minimum of 5 mg per week), or B cell depleting agents within the past 18 months (such as rituximab, ocrelizumab, or ofatumumab).
  - a. If taking MMF/MPA or MTX, the participant must have initiated therapy at least 8 weeks prior to randomization and be taking the same medications (regardless of dose) as at the time of the initial COVID-19 vaccine regimen. Note: Participants who withheld their IS medications around their initial vaccinations are eligible to participate.


- If enrolling in the B cell depleting therapy cohort, participant must have received an anti-CD20 or an anti-CD19 B cell depleting therapy in the past 18 months.
- 6. No changes in background IS medications, including MMF/MPA or MTX, in the 8 weeks prior to Screening, excluding the following:
  - a. HCQ,
  - b. Intraarticular steroids.
  - c. The addition of prednisone at ≤10mg per day or prednisone at any dose when given for ≤3 days, and
  - d. Corticosteroid bursts for non-autoimmune disease-related conditions, such as asthma or COPD, are permitted

#### **Exclusion Criteria:**

Individuals who meet any of these criteria are not eligible for randomization/allocation as study participants:

- 1. Inability or unwillingness of a participant to give assent or of a parent/guardian to give written informed consent, or of either to comply with study protocol.
- 2. History of severe allergic reaction to the initial COVID-19 vaccine regimen, or any component of any of the COVID-19 vaccines, or to PEG.
- 3. New diagnosis of malignancy that will require chemotherapy or immunotherapy, or ongoing treatment for a malignancy with chemotherapy or immunotherapy.
- 4. Active disease (per the Investigator's decision) resulting in inability to hold the IS therapy in the MMF/MPA or MTX arms of the study.
  - The potential impact of temporarily holding medication for participants with a recent mild disease flare within 4 weeks should be carefully considered.
- 5. Active disease during the Screening period resulting in:
  - a. an increase/addition of any IS medications, or
  - b. a suggestion of MS relapse per the investigator
- 6. Recent or current SARS-CoV-2 infection defined as:
  - a. Documented SARS-CoV-2 infection in the past 30 days (from the day the participant is diagnosed by positive test to Screening).
  - b. Positive result on a molecular COVID-19 test at Screening.
- 7. Receipt of a COVID-19 vaccine booster prior to Screening.
- Inflammatory myocarditis/pericarditis following initial COVID-19 vaccine regimen.

- Participants with active, ongoing chronic infections, including participants with evidence of:
  - a. HIV.
  - b. Hepatitis B as indicated by surface antigen.
  - c. Hepatitis C as indicated by anti-hepatitis C antibody positivity; if a participant is Hepatitis C antibody positive, they will be eligible to participate in the study if he/she is negative for viral load at Screening.

<u>Note:</u> Participants <u>are permitted to be on chronic prophylactic antimicrobial</u> <u>therapy.</u>

- Participants with common variable immunodeficiency disease, as well as any participants currently receiving immune globulin replacement therapy.
- 11. Participants who received licensed or investigational monoclonal antibodies or plasma products directed against SARS-CoV-2 within 30 days of Screening.
- 12. Participants who have received any live vaccines within 2 months of the anticipated study vaccine dose or who will have need of a live vaccine at any time during the study.
- 13. Currently pregnant or breastfeeding (postmenarchal females must have a negative urine pregnancy test at Screening)
- 14. Hemoglobin (Hgb) <8.0 g/dL (80 g/L)
- 15. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.
- 16. Other investigational chemical agent within 30 days or other investigational biologic agent within 8 weeks or 5 half-lives (whichever is longer) of Screening.
- 17. Concurrent treatment with cyclophosphamide.
- 18. Participants currently on any type of dialysis, or who have received a solid organ transplant.
- 19. Prisoners or participants who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be allowed to participant in this study.
- 20. Taking both MMF/MPA and MTX.
- Other investigational B cell depleting therapy as part of a clinical trial within 18
  months of Screening, unless drug assignment is known and the participant received
  an anti-CD20 or CD19 drug.
- 22. Participants with active systemic infections who have received systemic antimicrobials within the 14 days prior to Screening.


#### Study Stopping Rules

0BIf any of the events listed below occur, the DSMB chair will be notified, and a review of safety data will be performed to determine if enrollment in the study,

randomization/allocation, and/or administration of investigational study medication should be halted. If two weeks has elapsed and the DSMB has not met, then no new participants will be consented, allocated or randomized until after the DSMB completes review of the safety data.

#### Adult Participants:

Any of the following adverse events in adult participants attributable to the vaccine will trigger an *ad hoc* DSMB Safety Review:

- Death related to vaccine.
- Life-threating adverse event (Grade 4) related to vaccine.
- Permanent or severe disability related to vaccine.
- Occurrence of a Grade 3 or higher, vaccine-related SAE of the same type in 3 or more of the study participants who have received a study treatment. Note: Only SAEs occurring between Day 1 and the Week 24 study visit will be counted.
- Occurrence of severe flare or relapse after an additional homologous COVID-19 vaccine dose given at Stage 1, defined as within 12 weeks of the Stage Baseline/Week 0 visit (vaccination), in 3 of the first 10 participants or 30% thereafter, defined as follows.
- Occurrence of severe flare or relapse after a subsequent alternative COVID-19 vaccine dose given at Stage 2, defined as within 12 weeks of the Stage 2
  Baseline/Week 0 visit (vaccination), in 3 of the first 10 participants or 30% thereafter.

#### Pediatric Participants:

Any of the following adverse events in pediatric participants attributable to the vaccine will trigger an *ad hoc* DSMB Safety Review:

- Death related to vaccine
- Life-threatening AE (Grade 4) related to vaccine
- Permanent or severe disability related to vaccine
- Occurrence of a Grade 3 or higher, vaccine-related SAE of the same type in 3 or more of the study participants who have received a study treatment. Note: Only SAEs occurring between Day 1 and the Week 24 study visit will be counted.
- Occurrence of severe flare or relapse, between Baseline/Week 0 (vaccination) and the Week 12 visit, in 3 of the first 10 participants or 30% thereafter.

#### 4. GENERAL ANALYSIS AND REPORTING CONVENTIONS

The following is a list of general analysis and reporting conventions to be applied for this study:

- Categorical variables will be summarized using counts (n) and percents (%) and will be presented in the form n (%).
- Moment statistics including mean will be reported at 1 more significant digit than the
  precision of the original data. The standard deviation will be reported at 2 more
  significant digits than the precision of the original data. The level of precision may be
  modified on specific displays based on clinical judgement.
- Order statistics including median, min, and max will be reported to the same level of
  precision as the original observations. If any values are calculated to have more
  significant digits, then the value should be rounded so that it is the same level of
  precision as the original data.
- Following SAS default rules, the median will be reported as the average of the two
  middle numbers if the dataset contains an even number of observations.
- Test statistics including t and z test statistics will be reported to two decimal places.
- P-values will be reported to 3 decimal places if greater than 0.001; if less than 0.001, then
  they will be reported as '<0.001'. P-values and significant levels will be reported as 0.05
  rather than .05. A p-value will be reported as "1.000" only if it is exactly 1.000 without
  rounding. A p-value will be reported as "0.000" only if it is exactly 0.000 without
  rounding.</li>
- No preliminary rounding should be performed; rounding should only occur after analysis.
   To round, consider the digit to the right of last significant digit; if <5 then round down, and if ≥5 then round up.</li>
- In general, listings will be displayed by treatment arm and subject and will be sorted in the order that columns are displayed, starting with the first column on the left.
- All analyses will be performed using the SAS System version 9.4 or higher.


Version: 1.0

#### 5. ANALYSIS SAMPLES

Analysis samples for ACV01 for each study stage (Stage 1, Stage 2) and age group (Adult, Pediatric) will be defined as follows:

- Vaccinated population: will be defined as all participants who are randomized or allocated and receive study vaccine in the study. For all endpoints, participants will be evaluated by the actual vaccine received. In Cohorts A and B, participants will be analyzed in subgroups defined by randomized assignment to continue or withhold IS medications in the primary analysis.
- **Per protocol populations**: will be defined as the subgroup of participants in the vaccinated population who adhere to the treatment plan for IS medications defined in Section 7.1.1 Protocol-mandated Medications and have no major protocol deviations or ineligible entry criteria that would impact the vaccine response assessment at Week 4.
- **Safety population**: will be defined as all participants who initiate the treatment plan for IS medications or receive an additional dose of vaccine.

Document Control No.: TMP-SA-008-01 Template Effective Date: 23 Mar 2021

## 6. STUDY SUBJECTS

## 6.1. Disposition of Subjects

The disposition of participants will be summarized in tables and listed for each study stage (Stage 1, Stage 2) and age group (Adult, Pediatric). A CONSORT diagram outlining the flow of participants in the study will also be created. The numbers and percentages of participants randomized/allocated, in each analysis sample, and receiving vaccine, as well as reasons for early termination from the study, will be presented. For participants who were randomized/allocated but did not receive an additional dose of vaccine, the reasons for not receiving vaccine will also be presented. For Stage 2 of the study, the numbers and percentages of participants who are newly recruited vs. rollovers from Stage 1 will be summarized. Study disposition will also be summarized by site.

## 6.2. Demographic and Other Baseline Characteristics

Summary descriptive statistics for baseline and demographic characteristics will be reported for all analysis samples by study arm. Characteristics to be summarized include:

- Age, race, ethnicity, sex, body weight at screening, height
- Disease type and duration
- Roche Elecsys® Anti-SARS-CoV-2 S result at screening; both as a continuous variable and categorical: negative (≤0.79 U/mL) vs. positive (>0.79 U/mL); additionally, categorized as ≤0.79 U/mL, >0.79 U/mL through 50 U/mL, >50 U/mL through 200 U/mL, >200 U/mL
- History of prior SARS-CoV-2 infection at Screening
- Time (in weeks) from previous vaccine series
- Additional IS medications
- Steroid dose
- For Stage 2: previous vaccine series
- Medication dose for or Cohort A: MMF or MPA and Cohort B: MTX
- For Cohort C and Cohort F: B cell depletion therapy:
  - o Type of B cell depletion therapy
  - o Time (in weeks) from last dose of b cell depletion therapy to vaccine.
  - o CD19+B cells

#### 6.3. Prior and Concomitant Medications

Medications will be coded according to the World Health Organization (WHO) Drug Dictionary: WHO-Drug Global v2021-March. Medications will be reported on both the <u>Immunosuppressive</u> <u>Medication</u> and <u>Concomitant Medications</u> case report forms (CRFs).

The number and percentage of participants receiving IS medications will be presented overall and by medication class. Immunosuppressive medications will also be summarized by disease type. When reporting the number of subjects receiving the medication, a subject will only be counted once if they ever received the medication within the medication class. Percentages will be based on the number of subjects in the analysis population. Medications will also be listed.

The numbers and percentages of participants receiving the following concomitant medications will be presented overall and by medication class:

- SARS-CoV-2 vaccines or live vaccines (of any kind) administered outside of the study.
- Monoclonal antibodies administered for (a) pre-exposure prevention of COVID-19, (b) post-exposure prevention of COVID-19, or (c) treatment of COVID-19 infection.

## 6.4. Medical History

Analysis details will be provided in subsequent versions of the SAP.

#### 7. STUDY OPERATIONS

#### 7.1. Protocol Deviations

Protocol deviations will be listed by site with information such as date of deviation, category, description and reason for deviation, and corrective action taken. Protocol deviations will be summarized overall and by site in tabular format by type of deviation.

#### 7.2. Randomization and Allocation

When employed in any population, randomization will be accomplished through a password-protected, web-based randomization system. The investigators, clinic personnel, and participants will not be blinded to randomized treatment assignments. Statistical and project staff at the Statistical and Clinical Coordinating Center (SACCC) and the DAIT Medical Monitor and Project Manager will be unblinded to individual treatment assignments as well. Laboratories performing assays for this protocol will be blinded to the identity and group assignment of biological materials to be studied.

#### **7.2.1.** Adult Stage 1

Participants who sign the informed consent form and meet all eligibility criteria for Stage 1 will be assigned to cohorts defined by IS medication and by the initial COVID-19 vaccine regimen received. Participants in Cohort C will be allocated to continuing to take their prescribed IS medications throughout the trial. Participants in Cohorts A and B will be randomized in a balanced fashion (1:1), within the cohorts defined by IS medication and initial COVID-19 vaccine regimen, to one of the available IS medication treatment plans (continue cohort-defining IS vs. withhold cohort-defining IS). Randomization will be performed using a permuted block design stratified by disease type.

A total of 60 participants with a Roche Elecsys® Anti-SARS-CoV-2 S result ≤200 U/mL will be randomized or allocated to each arm. In each arm, the number of participants with Roche Elecsys® Anti-SARS-CoV-2 S results ≤50 U/mL will be capped at 40 participants, and the number of participants with Roche Elecsys® Anti-SARS-CoV-2 S results >50 U/mL and ≤200 U/mL will be capped at 40 participants.

## 7.2.2. Adult Stage 2

Participants who have signed the informed consent form and meet all eligibility criteria for Stage 2 will be allocated to cohorts defined by IS medication and by the initial COVID-19 vaccine regimen received. Participants who received either the Moderna COVID-19 Vaccine or Pfizer-BioNTech COVID-19 Vaccine will be allocated to the Stage 2 Arm that corresponds to their choice of either the Janssen vector-based COVID-19 vaccine or the other mRNA COVID-19 vaccine. Participants who received the Janssen COVID-19 Vaccine will be allocated to the Stage 2 Arm that corresponds to the Moderna COVID-19 Vaccine. Participants in Cohort D will withhold their MMF/MPA, participants in Cohort E will withhold their MTX, and any participants in Cohort F (B cell depletion therapy) who are also taking MMF/MPA or MTX will withhold these medications. No randomization will be employed.


A total of 60 participants with a Roche Elecsys® Anti-SARS-CoV-2 S result ≤200 U/mL will be allocated to each arm. In each arm, the number of participants with Roche Elecsys® Anti-SARS-CoV-2 S results ≤50 U/mL will be capped at 40 participants, and the number of participants with Roche Elecsys® Anti-SARS-CoV-2 S results >50 U/mL and ≤200 U/mL will be capped at 40 participants.

#### 7.2.3. Pediatric Population

Participants and their legal guardian(s) who sign the consent and assent forms, as appropriate to age, and meet all eligibility criteria for the pediatric portion of the trial will be assigned to cohorts defined by IS medication and by the initial COVID-19 vaccine regimen received. Participants in Cohort C will be allocated to continuing to take their prescribed IS medications throughout the trial. Participants in Cohorts A and B will be randomized in a balanced fashion (1:1), within the cohorts defined by IS medication and initial COVID-19 vaccine regimen, to one of the available IS medication treatment plans (continue IS vs. withhold IS). Randomization will be performed using a permuted block design stratified by disease type.

A total of 60 participants with a Roche Elecsys® Anti-SARS-CoV-2 S result ≤200 U/mL will be randomized or allocated to each arm. In each arm, the number of participants with Roche Elecsys® Anti-SARS-CoV-2 S results ≤50 U/mL will be capped at 40 participants, and the number of participants with Roche Elecsys® Anti-SARS-CoV-2 S results >50 U/mL and ≤200 U/mL will be capped at 40 participants.

## 7.3. Measures of Treatment Compliance

The number of participants who receive study vaccine will be summarized by arm.

In study arms that withhold IS medications around the time of vaccination, the total number of days, the number of days prior to vaccine, and the number of days post-vaccine that IS medications are withheld will be summarized.


Version: 1.0

#### 8. ENDPOINT EVALUATION

## 8.1. Overview of Efficacy Analysis Methods

#### 8.1.1. Multicenter Studies

Study participants will be recruited from 15-20 study sites for each of the adult and pediatric groups. Study data will be analyzed as a whole, and no formal accommodation for site-to-site variation will be made.

#### 8.1.2. Assessment Time Windows

Additional details will be provided in subsequent versions of the SAP.

#### 8.1.3. Timing of Analyses

The primary analysis will be evaluated independently within each arm (defined by age, cohort, vaccine, and IS treatment plan) in the vaccinated population, and will be conducted overall, in all participants with a Roche Elecsys® Anti-SARS-CoV-2 S result ≤200 U/mL at the Screening visit, and in the subgroup of participants with a Roche Elecsys® Anti-SARS-CoV-2 S result ≤50 U/mL at the Screening visit. Each analysis will occur after the evaluable participants assigned to that arm have completed the Week 4 study visit or are withdrawn from the study.

## 8.1.4. Multiple Comparisons/Multiplicity

The primary analysis will be evaluated independently within each arm, and p-values will not be adjusted for multiple comparisons.

All secondary analyses will be conducted in an exploratory fashion, with any p-values and confidence intervals presented as descriptive statistics with no adjustments for multiple comparisons.

## 8.2. Primary Endpoint

The primary endpoint of a protective antibody response will be the proportion of participants who reach the laboratory-defined threshold for the NIAID-VRC MSD 3 plex (Wu-1 full-length spike, RBD, and N proteins) assay at Week 4. The Wu-1 full-length spike protein will be used in determining a protective antibody response in the primary analysis; the RBD protein will be used in secondary analyses of antibody response; and N proteins will be used in supportive analyses as evidence of COVID infection.

## 8.2.1. Computation of the Primary Endpoint

The proportion of participants who reach the laboratory-defined threshold for the NIAID-VRC MSD 3 plex assay at Week 4 will be summarized by arm overall, in all participants with a Roche Elecsys® Anti-SARS-CoV-2 S result ≤200 U/mL at the Screening visit, and in the subgroup of participants with a Roche Elecsys® Anti-SARS-CoV-2 S result ≤50 U/mL at the Screening visit.


For concentrations that are below the Lower Limit of Detection (LLOD), numeric values equivalent to LLOD/2 are assigned before and for all descriptive reporting. Concentrations that are above the Upper Limit of Quantification are reported without adjustments.

Participants with missing Week 4 anti-COVID-19 antibody response data with a documented COVID infection prior to Week 4 will be considered as not having a protective antibody response. All other participants missing Week 4 anti-COVID-19 antibody response data will be considered to be missing-completely-at-random (MCAR).

### 8.2.2. Primary Analysis of the Primary Endpoint

The primary analysis will be evaluated independently within each arm (defined by stage, age, cohort, vaccine, and IS treatment plan) in the vaccinated population. The proportion of participants meeting a protective antibody response criteria will be reported in each arm with 90% Clopper-Pearson confidence intervals and analyzed using a one-sided exact test with alpha = 0.05 against the null hypothesis that the probability of achieving a protective immune response is  $\leq 0.25$ . P-values will not be adjusted for multiple comparisons.

The primary analysis will be conducted in all participants with a Roche Elecsys® Anti-SARS-CoV-2 S result ≤200 U/mL at the Screening visit, and in the subgroup of participants with a Roche Elecsys® Anti-SARS-CoV-2 S result ≤50 U/mL at the Screening visit. Each analysis will occur after the evaluable participants assigned to that arm have completed the Week 4 study visit or are withdrawn from the study.

### 8.2.3. Sensitivity Analyses of the Primary Analysis

A sensitivity analysis will be performed on the per protocol population.

### 8.2.4. Secondary Analyses of the Primary Endpoint

Descriptive statistics will be used to summarize antibody response to the additional homologous vaccine dose on a continuous scale, including median, minimum, and maximum, interquartile range, geometric mean, CV of the geometric mean, and 95% confidence intervals. Summary statistics, including 25th percentile, mean, median, and 75th percentile, will be plotted for each visit by treatment arm. Geometric mean and CV of the geometric mean will be computed as follows:

Geometric mean =  $\exp(\text{mean on log}_e \text{ scale})$ .

%CV geometric mean = 
$$\sqrt{\exp((SD \ on \ log_e \ scale)^2) - 1} \ x \ 100$$

Primary and secondary analyses will be repeated for the RBD proteins to summarize antibody response to the additional homologous vaccine dose on a continuous scale. Supportive analyses will use descriptive statistics to summarize N protein levels as evidence of COVID infection.

In the final analysis, supportive analyses will also use a multivariable regression model on the entire vaccinated population in order to estimate the rates of vaccine response within and across arms (age group, cohort, vaccine, and IS treatment plan group) using the logistic link function, and including baseline covariates for disease type (SLE, RA, MS, SSc, and pemphigus in adults


and JIA, pediatric SLE, JDM, and POMS in pediatrics) and immune response to the initial COVID-19 vaccine regimen (anti-COVID-19 antibody negative or positive).

Estimates of the average antibody response and variance within and across cohorts will be obtained from a multivariate general linear regression model. Based on published data on the assays, it is anticipated that log-transformation of assay values will allow for Gaussian assumptions to hold, but alternative Box-Cox transformations of the data may be explored to stabilize the variance.

The primary and supportive analyses will also be replicated on the Per protocol population and using alternative strategies for missing data. Additional analysis details will be provided in subsequent versions of the SAP.

### 8.3. Secondary Endpoints

#### 8.3.1. Seroconversion at Week 4

Seroconversion at Week 4, following additional doses of COVID-19 vaccine, will be assessed in the subgroup of participants in the vaccinated population that are anti-COVID-19 antibody negative at Week 0. Seroconversion will be assessed separately with (a) the NIAID-VRC MSD 3 plex assay and (b) the Roche Elecsys® Anti-SARS-CoV-2 S electrochemiluminescence immunoassay.

The subgroup of participants that are anti-COVID-19 antibody negative at Week 0 will be defined as having a result less than or equal to the positive threshold value listed below at the Week 0/Baseline visit.

Seroconversion will be defined as a having a result greater than the positive threshold value listed below at the Week 4 visit. Seroconversion will be defined in a similar fashion for subsequent follow-up visits through Week 48 as well. Participants with missing anti-COVID-19 antibody response data will be considered to be MCAR.

The following positive thresholds will be used:

| | | Positive |
|---|---|---|
| Assay | Test | Threshold |
| NIAID-VRC MSD 3 plex | Wu-1 full-length spike | 1,204.71 AU/mL |
| NIAID-VRC MSD 3 plex | RBD | 517.86 AU/mL |
| Roche Elecsys® Anti-SARS-CoV-2 S | COVID-19 Spike | 0.70 II/mI |
| electrochemiluminescence immunoassay | Domain Antibody | 0.79 U/mL |

The proportions who seroconvert within arms will be summarized using 95% Clopper-Pearson confidence intervals in preliminary analyses. In the final analysis, comparisons of rates of seroconversion across arms and subgroups will use a two-sample Binomial exact test with nominal two-sided alpha = 0.05.

Supportive analyses will evaluate seroconversion of N protein levels in the NIAID-VRC MSD 3 plex assay (Threshold = 9,779.62 AU/ml) as evidence of COVID infection.


### 8.3.2. Fold Increase in anti-COVID-19 Antibody Levels at Week 4

Fold increase in anti-COVID-19 antibody levels will be assessed for the subgroups of participants in the vaccinated population that are anti-COVID-19 antibody positive at Week 0 using separately (a) the NIAID-VRC MSD 3 plex assay and (b) the Roche Elecsys® Anti-SARS-CoV-2 S electrochemiluminescence immunoassay.

The subgroup of participants that are anti-COVID-19 antibody positive at Week 0 will be defined as having a result greater than the positive threshold value listed below at the Week 0/Baseline visit.

The following positive thresholds will be used:

| | | Positive |
|---|---|---|
| Assay | Test | Threshold |
| NIAID-VRC MSD 3 plex | Wu-1 full-length spike | 1,204.71 AU/mL |
| NIAID-VRC MSD 3 plex | RBD | 517.86 AU/mL |
| Roche Elecsys® Anti-SARS-CoV-2 S | COVID-19 Spike | 0.79 U/mL |
| electrochemiluminescence immunoassay | Domain Antibody | 0.79 U/IIIL |

Participants with missing anti-COVID-19 antibody response data will not be imputed.

Fold improvement for each assay will be defined as follows and will be defined in a similar fashion for subsequent follow-up visits through Week 48 as well:

$$Fold\ improvement = \frac{anti\text{-COVID-19 Antibody Response}_{\text{Week 4}}}{anti\text{-COVID-19 Antibody Response}_{\text{Baseline}}}$$

Descriptive statistics will be used to summarize fold increase in anti-COVID-19 antibody levels at Week 4, including median, minimum, and maximum, geometric mean, CV of the geometric mean, and 95% confidence intervals.

Supportive analyses will evaluate fold increase in N protein levels in the NIAID-VRC MSD 3 plex assay (Threshold = 9,779.62 AU/ml) as evidence of COVID infection.

### 8.3.3. Longitudinal Changes in anti-COVID-19 Antibody Responses

Longitudinal changes in anti-COVID-19 antibody responses will be analyzed from Week 0 to Weeks 4, 12, 24, 36, and 48 and will be summarized over time by study visit using descriptive statistics. This endpoint will not be evaluated in preliminary analyses. Additional analysis details will be provided in subsequent versions of the SAP.

### 8.3.4. Longitudinal Changes in Neutralization and Pseudo Neutralization Assays

Longitudinal changes in neutralization and pseudo neutralization assays will be assessed from Week 0 to Weeks 4, 12, 24, 36, and 48 and will be summarized by study visit using descriptive statistics. This endpoint will not be evaluated in preliminary analyses. Additional analysis details will be provided in subsequent versions of the SAP.


### 8.3.5. Changes in Diseases Activity using CGI-C

Changes in disease activity after receipt of additional doses of COVID-19 vaccine will be assessed as measured by the CGI-C. In preliminary analyses, the change in CGI-C from Week 0 to Week 4 will be summarized in each study population using descriptive statistics. Analysis details will be provided in subsequent versions of the SAP.

### 8.3.6. Changes in Diseases Activity using PGA

Changes in disease activity after receipt of additional doses of COVID-19 vaccine will be assessed as measured by the PGA. This endpoint will not be evaluated in preliminary analyses. Analysis details will be provided in subsequent versions of the SAP.

### 8.3.7. Changes in Disease Activity as Measured by Disease-Specific Assessments

Longitudinal changes in disease activity will not be evaluated in preliminary analyses. The proportion of participants who meet the definition for disease-specific flares by Week 4 will be summarized in preliminary analyses.

### 8.3.7.1. H-SLEDAI and SELENA-SLEDAI Flare Index

Disease activity for SLE participants will be measured by the (H-SLEDAI and SELENA-SLEDAI Flare Index for SLE. Analysis details will be provided in subsequent versions of the SAP.

#### 8.3.7.2. DAS28-CRP

Disease activity for RA participants will be measured by the DAS28-CRP for RA. Analysis details will be provided in subsequent versions of the SAP.

### 8.3.7.3. Flare assessment for SSc

Disease activity for SSc participants will be measured using the flare assessment for SSc (including patient-reported flare assessment). Analysis details will be provided in subsequent versions of the SAP.

### 8.3.7.4. PDAI

Disease activity for pemphigus participants will be measured using the PDAI for pemphigus. Analysis details will be provided in subsequent versions of the SAP.

### 8.3.7.5. Physician-assessed relapse for MS

Disease activity for MS participants will be measured using the physician-assessed relapse for MS. Analysis details will be provided in subsequent versions of the SAP.

### 8.3.7.6. JADAS-10

Disease activity for JIA participants will be measured using the JADAS-10 for polyarthritis, enthesitis related to JIA, oligoarthritis, and psoriatic arthritis. Analysis details will be provided in subsequent versions of the SAP.

#### 8.3.7.7. PASI

Disease activity for JIA participants will also be measured using the PASI for psoriatic arthritis. Analysis details will be provided in subsequent versions of the SAP.

#### 8.3.7.8. SLEDAI-2K and Childhood-onset SLE Criteria for Global Flare

Disease activity for pediatric SLE will be measured using the SLEDAI-2K and Childhood-onset SLE Criteria for Global Flare [1] for pediatric SLE. Analysis details will be provided in subsequent versions of the SAP.

### 8.3.7.9. CMAS

Disease activity for JDM will be measured using the CMAS for JDM. Analysis details will be provided in subsequent versions of the SAP.

#### 8.3.7.10. JDM DAS

Disease activity for JDM will be measured using the JDM DAS for JDM. Analysis details will be provided in subsequent versions of the SAP.

### 8.3.7.11. Physician-assessed relapse for POMS

Disease activity for POMS will be measured using the physician-assessed relapse for MS for POMS. Analysis details will be provided in subsequent versions of the SAP.

### 8.3.8. Changes in Patient-reported Outcomes

#### 8.3.8.1. PROMIS 29

Changes in the PROMIS 29 will be assessed in the adult population. Analysis details will be provided in subsequent versions of the SAP.

### 8.3.8.2. **PedsQL**

Changes in the PedsQL will be assessed in the pediatric population. Analysis details will be provided in subsequent versions of the SAP.

### 8.3.8.3. PtGA

Changes in the PtGA will be assessed in the adult and pediatric populations. Analysis details will be provided in subsequent versions of the SAP.

The National Institute of Allergy and Infectious Diseases (NIAID) Statistical Analysis Plan - Protocol ACV01

### 8.3.8.4. PGI-C

Changes in the PGI-C will be assessed in the adult and pediatric populations. Analysis details will be provided in subsequent versions of the SAP.

### 8.4. Other Endpoints

Analysis details will be provided in subsequent versions of the SAP.

### 8.5. Examination of Subgroups

Analysis details will be provided in subsequent versions of the SAP.

### 9. SAFETY EVALUATION

### 9.1. Overview of Safety Analysis Methods

All safety analyses will be carried out using the safety sample defined in Section 5 unless otherwise noted. Missing safety information will not be imputed. These analyses will not be stratified by site.

### 9.2. Adverse Events

For this study, solicited AEs are predefined local and systemic events for which the participants will be specifically questioned, and which will be noted by these participants. An AE is considered "unsolicited" when it is collected through an open-ended question and is not specified as a solicited AE. An MAAE is defined as a hospitalization, emergency room visit, or an otherwise unscheduled visit to or from medical personnel for any reason; and considered related to study vaccine. A NOCMC is defined as any new ICD diagnosis (per current International Statistical Classification of Diseases and Related Health Problems) that is applied to the study participant during the course of the study, after receipt of the vaccine, that is expected to continue for at least 3 months and requires continued health care intervention. An AE is considered "serious" if, in the view of either the investigator or Sponsor (DAIT/NIAID), it results in any of the following outcomes: death, life-threatening, hospitalization, persistent or significant incapacity, congenital anomaly or birth defect, or is considered an important medical event. See protocol Section 12.2 for more details on AE definitions.

The collection periods and reporting for AEs are as follows:

- Solicited AEs (all grades) will be collected from Day 1 (vaccine administration) through 7 days post study vaccination using the MyOwnMed vaccine reaction diary.
  - Investigators are responsible for reporting solicited AEs in the electronic data capture system (EDC) in the following special cases:
    - If a solicited AE is also an SAE or MAAE must be entered in EDC to capture additional information about the event.
    - If a solicited AE, previously reported in MyOwnMed, is found to be ongoing at Day 7 (post vaccination), the solicited AE must be entered in EDC so it can be followed to resolution, with or without sequelae.
    - Unsolicited AEs (unrelated to reactogenicity) that are entered into the Vaccine Reaction Diary and are also identified during the Week 1 visit are to be reported in EDC
- Unsolicited AEs will be collected as follows and reported in EDC:
  - Any unsolicited AEs that are Grade 3 or higher will be collected from randomization/allocation through vaccination administration.
  - o All unsolicited AEs (all grades) will be collected from Day 1 through Day 28.


- Any flares of a secondary autoimmune disease will be reported as an unsolicited AE (all grades) and will be collected from Day 1 through the end of the participant's study participation.
- SAEs, MAAEs, and NOCMCs will be collected from Day 1 through the end of the
  participant's study participation, regardless of the National Cancer Institute's (NCI's)
  Common Toxicity Criteria for Adverse Events (CTCAE) grade, and reported in EDC.
- COVID-19 diagnoses (all grades) confirmed by molecular COVID-19 testing will be collected from Day 1 through the end of the participant's study participation and reported in EDC.

All AEs will be classified by system organ class (SOC) and preferred term, according to a standardized thesaurus (Medical Dictionary for Regulatory Activities [MedDRA] version 24.0).

Grading criteria are defined as follows:

- Solicited AEs: Participants will grade solicited AEs using a 0-3 (no symptom, mild, moderate, and severe) participant symptom rating scale as outlined in the Vaccine Reaction Diary instructions.
- Allergic reactions: The investigator will grade severity of systemic allergic reactions on a scale of 1 to 5 according to criteria set forth in the Consortium of Food Allergy Research (CoFAR) Grading Scale modified for use in adults only (See Protocol Section 20.2 CoFAR Grading Scale for Systemic Allergic Reactions Version 3.0).
- Liver Function Abnormalities: Liver function abnormalities will be graded using alternative criteria, which are based on the NCI-CTCAE version 4.0, and are defined relative to the upper limit of normal (ULN) as defined in Protocol Section 12.3.1 *Grading Criteria*.
- All other events: The study site will grade the severity of all other AEs experienced by
  the study participants according to the criteria set forth in the NCI-CTCAE version 5.0 as
  deemed appropriate for the 5 adult autoimmune diseases and 4 pediatric autoimmune
  diseases, and use of background IS medications of interest in this trial.

If the start date of an AE is incomplete or missing, it will be assumed to have occurred on or after the first dose of investigational product, except if an incomplete date (e.g., month and year) clearly indicates that the event started prior to treatment

If a subject experiences the same AE on multiple occasions, the event will be counted once for each occurrence when reporting the number of AEs. When reporting the number of subjects experiencing the events, a subject will only be counted once if they experience at least one event within the particular SOC or preferred term. Percentages will be based on the number of subjects in the safety population. The tabular summaries will be sorted by descending frequency by SOC and preferred term (PT) in the treatment group arm.

Summary tables will be reported for treatment emergent adverse events unless otherwise indicated. An overall summary table will include:


- Total number of events, and number and percentage of subjects experiencing at least one event for the following categories:
  - AEs
  - SAEs
  - AEs related to study vaccine
  - AE leading to study vaccine discontinuation
  - AE leading to death
  - MAAEs
  - NOCMCs
  - SARS-CoV-2 infections
  - Solicited Adverse Events
  - AEs by severity

AEs classified by MedDRA SOC and preferred term will be summarized for each treatment group for each of the following:

- o All AEs
- All Related AEs
- o All SAEs
- All AEs leading to study drug discontinuation
- AEs by severity
- o AEs by relationship to study drug

Listings of all AEs, MAAEs, and NOCMCs will be provided for the safety population.

### 9.2.1. Solicited Adverse Events

Participants are provided access to an electronic 7-day diary to aid in recording solicited local and systemic reactions to the vaccine, as well as symptoms of a potential allergic reaction, unsolicited AEs, and concomitant medications, including start and stop dates. The diary includes instructions for participants on how to take an oral temperature and how to measure injection site reactions. A paper copy of the diary may be provided for participants who do not have a device to access the electronic diary or as a backup collection tool. A member of the study team will review the information in the diary with the participant, including how to use and access the electronic diary, and will record adverse events on the CRF page as appropriate based on review of the diary.

Summary displays based on the maximum severity of solicited symptoms reported over the 7-day period will be presented in tables and graphically by study arm. Summaries of the diary entries over the 7-day period will also be presented by study arm.

# 9.3. Deaths, Serious Adverse Events, and Other Significant Adverse Events

Serious AEs classified by MedDRA SOC and PT will be summarized for each treatment group and overall for each of the following:

• All serious AEs


The National Institute of Allergy and Infectious Diseases (NIAID) Statistical Analysis Plan - Protocol ACV01

- Serious AEs by severity
- Serious AEs by relationship to study drug

Rules for counting SAEs in summary tables are the same as those applied to AEs reported in Section 9.3.

All SAEs and SAEs resulting in death will be presented in data listings for subjects in the safety population. A separate display listing will be created for all deaths summarizing the time to death and cause of death.

### 9.4. Clinical Laboratory Evaluation

Analysis details will be provided in subsequent versions of the SAP.

# 9.5. Vital Signs, Physical Findings, and Other Observations Related to Safety

### 9.5.1. Vital Signs

Analysis details will be provided in subsequent versions of the SAP.

### 9.5.2. Physical Examinations

Analysis details will be provided in subsequent versions of the SAP.

### 9.5.3. Other Safety Measures

Analysis details will be provided in subsequent versions of the SAP.


Version: 1.0

The National Institute of Allergy and Infectious Diseases (NIAID) Statistical Analysis Plan - Protocol ACV01

### 10. OTHER ANALYSES

Analysis details will be provided in subsequent versions of the SAP.

### 11. INTERIM ANALYSES AND DATA MONITORING

The progress of the study will be monitored by the NIAID DSMB. The NIAID Autoimmune DSMB is chartered to review safety data and to make recommendations to NIAID regarding continuation, termination, or modification of the study. The DSMB will review the safety data within 6 months after the first participant is treated, and an initial review should occur no later than after this first arm has closed to enrollment and all participants completed 4 weeks of follow up. Following the initial review, the DSMB will review the safety data approximately every 6 months during planned DSMB Data Review Meetings. Data for the planned safety reviews will include, at a minimum, a listing of all reported AEs, SAEs, MAAEs, NOCMCs, and increases in autoimmune disease activity (flares/relapses).

The DSMB chair will be informed of any IND Safety Reports in a timely manner in order to make a recommendation for an ad hoc full board review and /or protocol suspension. In addition, safety data will be reviewed by the DSMB when an event occurs that is of sufficient concern to the NIAID medical monitor or protocol co-chairs to warrant review, or when an event occurs that could contribute to a stopping rule.

Document Control No.: TMP-SA-008-01 Template Effective Date: 23 Mar 2021

### 12. CHANGES TO THE ANALYSES PLANNED IN THE PROTOCOL

1. The protocol specifies that the analysis of primary and secondary endpoints will be evaluated independently within each arm (defined by age, cohort, vaccine, and IS treatment plan) and conducted in (1) all participants with a Roche Elecsys® Anti-SARS-CoV-2 S result ≤200 U/mL at the Screening visit, and (2) in the subgroup of participants with a Roche Elecsys® Anti-SARS-CoV-2 S result ≤50 U/mL at the Screening visit. Each analysis of the primary endpoint will occur after the evaluable participants assigned to that arm and subgroup have completed the Week 4 study visit or are withdrawn from the study. For the purposes of this document, we refer to analyses at this timepoint as preliminary, and a final analysis will occur once all participants have completed or withdrawn from the study.

If at the point of each preliminary analysis, a definition of a protective antibody response using a laboratory-defined threshold for responses within the NIAID-VRC MSD 3 plex assay is unavailable, the primary analysis of primary and secondary endpoints will not be performed, and only the secondary analysis to summarize antibody response on a continuous scale using descriptive statistics will be performed.

2. Protocol Section 13.4.4, *Analyses of Secondary and Other Endpoint(s)*, notes "The incidence of seroconversion following additional vaccine doses of COVID-19 vaccine will be evaluated in the subgroups of participants that are anti-COVID-19 antibody negative at baseline using separately, (a) NIAID-VRC MSD 3 plex (Wu-1 full-length spike, RBD, and N) assay with thresholds <1204.7 and 517.9 proteins AU/mL, respectively, and (b) the Roche Elecsys® Anti-SARS-CoV-2 S electrochemiluminescence immunoassay with a threshold <0.80 U/mL." Seroconversion will not be assessed using the N proteins test as it is a measure of natural infection rather than vaccine response.


Version: 1.0

The National Institute of Allergy and Infectious Diseases (NIAID) Statistical Analysis Plan - Protocol ACV01

### 13. REFERENCES

NA.

### 14. APPENDIX

### 14.1. Study Flow Chart

Figure 1. Participant Flow Diagram for Adult Stage 1

Stage 1: Additional Homologous Vaccine



IS = immunosuppressive medications; MMF = mycophenolate mofetil; MPA = mycophenolic acid; MS = multiple sclerosis; MTX = methotrexate; RA = rheumatoid arthritis; SLE = systemic lupus erythematosus; SSc = systemic sclerosis

Figure 2. Study Flow for Adult Stage 1



IS = immunosuppressive medication


Figure 3. Participant Flow Diagram for Adult Stage 2

### Stage 2: Additional alternative vaccine



IS = immunosuppressive medications; MMF = mycophenolate mofetil; MPA = mycophenolic acid; MS = multiple sclerosis; MTX = methotrexate; RA = rheumatoid arthritis; SLE = systemic lupus erythematosus; SSc = systemic sclerosis

Figure 4. Study Flow for Adult Stage 2



IS = immunosuppressive; MMF = mycophenolate mofetil; MPA = mycophenolic acid


<sup>\*</sup> Additional homologous vaccine dose is defined as a third dose of the Pfizer-BioNTech COVID-19 Vaccine or Moderna COVID-19 Vaccine, or a second dose of the Janssen COVID-19 Vaccine.

<sup>¥</sup> Pfizer-BioNTech COVID-19 Vaccine or Moderna COVID-19 Vaccine, whichever was not received for the initial regimen and additional homologous dose.

Figure 5. Participant Flow Diagram for Pediatric Participants

### Pediatric Additional Homologous Vaccine

Cohort A: MMF/MPA and Cohort B: MTX



IS = immunosuppressive medications; JDM = juvenile dermatomyositis; JIA = juvenile idiopathic arthritis; POMS = pediatriconset multiple sclerosis; MMF = mycophenolate mofetil; MPA = mycophenolic acid; MTX = methotrexate; SLE = systemic lupus erythematosus

Figure 6. Study Flow Diagram for Pediatric Participants



IS = immunosuppressive medication


<sup>\*</sup>Treatment arm will be opened for enrollment when authorization or approval of these vaccines is granted for the pediatric population(s).

The National Institute of Allergy and Infectious Diseases (NIAID) Statistical Analysis Plan - Protocol ACV01

### 14.2. Schedule of Events

See protocol Section 20.1, Schedules of Events, for more details.

The National Institute of Allergy and Infectious Diseases (NIAID) Statistical Analysis Plan - Protocol ACV01

### 15. ATTACHMENTS

NA.

# ACKNOWLEDGEMENT AND SIGNATURE SHEET

| Approved: | Approved: |
|---|---|
| Principal Biostatistician | Principal Statistical Scientist |
| Signature and Date | Signature and Date |
| DocuSigned by: Signing Reason: I approve this document Signing Time: 16-Mar-2022 10:43:23 PM EDT 284D7D99CF8C44E389ABAF99B28BBBE9 | DocuSigned by: Signing Reason: I approve this document Signing Time: 17-Mar-2022 11:06:53 AM EDT 4CF69AFD2FC0473D9FC0D9F733FFEA26 |

| Approved: | Approved: |
|---|---|
| Medical Monitor | Medical Monitor |
| Signature and Date | Signature and Date |
| DocuSigned by: Signing Reason: I approve this document Signing Time: 17-Mar-2022 9:29:34 AM EDT 765A331086DC4DF5AD2A6ACEC3FACD5E | DocuSigned by: Signing Reason: I approve this document Signing Time: 16-Mar-2022 5:22:35 PM EDT F516482134FC4FDDAF3288BD039F6ECC |

| Approved: | Approved: |
|---|---|
| Judith James, MD, PhD | Meggan Mackay, MD, MS |
| Protocol Co-Chair | Protocol Co-Chair |
| Signature and Date | Signature and Date |
| DocuSigned by: Julitle James | DocuSigned by: Meggan Mackay |
| Signer Name: Judith James Signing Reason: I approve this document Signing Time: 16-Mar-2022 2:14:19 PM EDT 01C3137148084E71A42CA9A2B9E2A802 | Signer Name: Meggan Mackay Signing Reason: I approve this document Signing Time: 17-Mar-2022 12:45:25 PM EDT 2464E5AFBC954423A68E6337D94689E5 |

| Approved: | Approved: |
|---|---|
| Dinesh Khanna, MBBS, MSC | Amit Bar-Or, MD, FRCPC |
| Protocol Co-Chair | Protocol Co-Chair |
| Signature and Date | Signature and Date |
| DocuSigned by: Direct Elanna Signer Name: Dinesh Khanna Signing Reason: I approve this document Signing Time: 16-Mar-2022 12:22:53 PM EDT 7C116CC28BE94B1BBCCBF7BF9FC92120 | |

| Approved: | Approved: |
|---|---|
| Virginia Pascual, MD | Stacy Ardoin, MD |
| Protocol Co-Chair | Protocol Co-Chair |
| Signature and Date | Signature and Date |
| DocuSigned by: | DocuSigned by: |
| Virginia Pascual Signer Name: Virginia Pascual Signing Reason: I approve this document Signing Time: 16-Mar-2022 12:23:47 PM EDT 600745241B59467B82ED5ED47F214D2D | Stary Irdoin Signer Name: Stacy Ardoin Signing Reason: I approve this document Signing Time: 20-Mar-2022 12:24:43 PM EDT 6695E7A3F92C4B1694DA1BFC14F98F68 |

| Approved: | Approved: |
|---|---|
| Natasha Mckerran Ruth, MD | Tracey Wright, MD |
| Protocol Co-Chair | Protocol Co-Chair |
| Signature and Date | Signature and Date |
| DocuSigned by: Natasha Mckerran Kuth Signer Name: Natasha Mckerran Ruth Signing Reason: I approve this document Signing Time: 16-Mar-2022 1:42:52 PM EDT | DocuSigned by: Tracy B. (Wright, MI) Signer Name: Tracey B. Wright, MD Signing Reason: I approve this document Signing Time: 16-Mar-2022 1:13:41 PM EDT |
| CDE71CEB76764AB4BD23AF440A9CEC2E | 7EFC6823A13941DCA79C34B24E62EFE5 |

### **Certificate Of Completion**

Envelope Id: 86FFBADB7591451298003B78F9D1424B

Subject: ACV01 SAP Signature

Source Envelope: Document Pages: 2

Certificate Pages: 8

AutoNav: Enabled **Envelopeld Stamping: Disabled** 

Time Zone: (UTC-05:00) Eastern Time (US & Canada)

Status: Completed

Envelope Originator:

2635 E NC Hwy 54 Durham, NC 27713

IP Address: 4.34.23.236

### **Record Tracking**

Status: Original

3/16/2022 11:57:58 AM

Security Appliance Status: Connected Storage Appliance Status: Connected

Holder:

Pool: FedRamp Pool: Rho, Inc.

Signatures: 11

Initials: 0

Location: DocuSign

Location: DocuSign

Sent: 3/16/2022 12:21:11 PM Viewed: 3/16/2022 10:39:40 PM Signed: 3/16/2022 10:43:29 PM

Sent: 3/16/2022 12:21:11 PM Viewed: 3/17/2022 11:06:33 AM Signed: 3/17/2022 11:07:28 AM

**Timestamp** 

#### Signer Events

Security Level: Email, Account Authentication (Required)



Signature Adoption: Pre-selected Style

284D7D99-CF8C-44E3-89AB-AF99B28BBBE9

Using IP Address: 4.34.23.236

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

#### Signature



Signature ID:

I approve this document

#### Electronic Record and Signature Disclosure: Not Offered via DocuSign





Security Level: Email, Account Authentication (Required)



Signature Adoption: Pre-selected Style

Signature ID:

4CF69AFD-2FC0-473D-9FC0-D9F733FFEA26

Using IP Address: 4.34.23.236

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

#### **Electronic Record and Signature Disclosure:** Not Offered via DocuSign

### Signer Events

Dinesh Khanna

khannad@med.umich.edu

Partner

Security Level: Email, Account Authentication (Required)

#### Signature

DocuSigned by:

Dinesh Elanna



Signer Name: Dinesh Khanna Signing Reason: I approve this document Signing Time: 16-Mar-2022 | 12:22:53 PM EDT -7C116CC28BE94B1BBCCBF7BF9FC92120 Timestamp

Sent: 3/16/2022 12:21:13 PM Viewed: 3/16/2022 12:22:37 PM Signed: 3/16/2022 12:22:58 PM

Signature Adoption: Pre-selected Style

Signature ID:

7C116CC2-8BE9-4B1B-BCCB-F7BF9FC92120

Using IP Address: 68.62.19.191

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document



Accepted: 3/16/2022 12:22:37 PM ID: b3fafcc8-9992-4ba5-9e90-2a3b3452d1f5



Sent: 3/16/2022 12:21:12 PM Viewed: 3/16/2022 5:15:33 PM Signed: 3/16/2022 5:22:41 PM

Security Level: Email, Account Authentication (Required)

Signature Adoption: Pre-selected Style

Signature ID:

F5164821-34FC-4FDD-AF32-88BD039F6ECC

Using IP Address: 128.231.234.68

With Signing Authentication via DocuSign password With Signing Reasons (on each tab):

I approve this document

#### Electronic Record and Signature Disclosure:

Accepted: 8/22/2020 3:45:44 PM ID: 5626e8be-940c-4427-b70c-5a067a412344



Sent: 3/16/2022 12:21:12 PM Viewed: 3/17/2022 9:28:52 AM Signed: 3/17/2022 9:29:47 AM

Security Level: Email, Account Authentication (Required)

Signature Adoption: Pre-selected Style

Signature ID:

765A3310-86DC-4DF5-AD2A-6ACEC3FACD5E

Using IP Address: 67.165.240.30

With Signing Authentication via DocuSign password With Signing Reasons (on each tab):

I approve this document

### Electronic Record and Signature Disclosure:

Accepted: 9/27/2020 8:50:43 PM ID: 30600a06-8cc9-47f3-9e24-5859ba13eafe

### **Signer Events**

**Judith James** 

Judith-James@omrf.org

Security Level: Email, Account Authentication (Required)

### Signature

—DocuSigned by: Juditle James

U

Signer Name: Judith James
Signing Reason: I approve this document
Signing Time: 16-Mar-2022 | 2:14:19 PM EDT

-01C3137148084E71A42CA9A2B9E2A802

Timestamp

Sent: 3/16/2022 12:21:14 PM Viewed: 3/16/2022 2:13:04 PM Signed: 3/16/2022 2:14:24 PM

Sent: 3/16/2022 12:21:14 PM

Resent: 3/17/2022 12:35:07 PM Viewed: 3/17/2022 12:45:00 PM

Signed: 3/17/2022 12:45:45 PM

Sent: 3/16/2022 12:21:15 PM

Viewed: 3/16/2022 1:42:20 PM Signed: 3/16/2022 1:43:02 PM

Signature Adoption: Pre-selected Style

Signature ID:

01C31371-4808-4E71-A42C-A9A2B9E2A802

Using IP Address: 156.110.145.246

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

#### Electronic Record and Signature Disclosure:

Accepted: 3/16/2022 2:13:04 PM ID: 8e4568ef-90b4-462d-8cc7-00c5b93ad4f8

Meggan Mackay

mmackay@northwell.edu

MD

Security Level: Email, Account Authentication

(Required)

### Meggan Mackay

Signature Adoption: Pre-selected Style

Signature ID:

2464E5AF-BC95-4423-A68E-6337D94689E5

Using IP Address: 69.27.229.130

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

### Electronic Record and Signature Disclosure:

Accepted: 12/3/2021 10:28:55 AM ID: a9f3ff03-031d-4ff7-930e-d639278d301f

Natasha Mckerran Ruth

ruthn@musc.edu

Security Level: Email, Account Authentication

(Required)

-DocuSigned by:

Nataslia McKerran Kutli

Signer Name: Natasha Mckerran Ruth Signing Reason: I approve this document Signing Time: 16-Mar-2022 | 1:42:52 PM EDT

-CDE71CEB76764AB4BD23AF440A9CEC2E

Signature Adoption: Pre-selected Style

Signature ID:

U

CDE71CEB-7676-4AB4-BD23-AF440A9CEC2E

Using IP Address: 76.23.125.236

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

### Electronic Record and Signature Disclosure:

Accepted: 3/16/2022 1:42:20 PM ID: e799f907-edc7-4fb5-a123-9d974d4c468c

| Signer Events | Signature | Timestamp |
|---|---|---|
| Stacy Ardoin stacy.ardoin@nationwidechildrens.org Security Level: Email, Account Authentication (Required) Electronic Record and Signature Disclosure: Accepted: 3/20/2022 12:24:02 PM | Stary Indian Signature Adoption: Pre-selected Style Signature ID: 6695E7A3-F92C-4B16-94DA-1BFC14F98F68 Using IP Address: 69.24.144.18 With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document | Sent: 3/16/2022 12:21:15 PM Resent: 3/17/2022 12:35:07 PM Viewed: 3/20/2022 12:24:02 PM Signed: 3/20/2022 12:24:50 PM |
| ID: 1e81ac1d-6965-4b21-a997-a3300d5a3f9d | | |
| Tracey B. Wright, MD tracey.wright@utsouthwestern.edu Security Level: Email, Account Authentication (Required) Electronic Record and Signature Disclosure: Accepted: 3/16/2022 1:12:08 PM ID: d91b8622-a08f-4f76-9280-e78d8d642f28 | DocuSigned by: Tracy B. (Wriph, ML) Signer Name: Tracey B. Wright, MD Signing Reason: I approve this document Signing Time: 16-Mar-2022 1:13:41 PM EDT 7EFC6823A13941DCA79C34B24E62EFE5 Signature Adoption: Pre-selected Style Signature ID: 7EFC6823-A139-41DC-A79C-34B24E62EFE5 Using IP Address: 129.112.109.53 With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document | Sent: 3/16/2022 12:21:16 PM<br>Viewed: 3/16/2022 1:12:08 PM<br>Signed: 3/16/2022 1:13:45 PM |
| Virginia Pascual | DocuSigned by: | Sent: 3/16/2022 12:21:16 PM |
| vip2021@med.cornell.edu | Virginia Pascual | Viewed: 3/16/2022 12:23:00 PM |
| MD<br>Security Level: Email, Account Authentication<br>(Required) | Signer Name: Virginia Pascual Signing Reason: I approve this document Signing Time: 16-Mar-2022 12:23:47 PM EDT 600745241B59467B82ED5ED47F214D2D | Signed: 3/16/2022 12:23:56 PM |
| Electronic Record and Signature Disclosure: Accepted: 3/16/2022 12:23:00 PM ID: ee99b2af-8977-42f1-8228-adeffb1ca95e | Signature Adoption: Pre-selected Style Signature ID: 60074524-1B59-467B-82ED-5ED47F214D2D Using IP Address: 96.224.244.124 With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document | |
| In Person Signer Events | Signature | Timestamp |
| Editor Delivery Events | Status | Timestamp |

Timestamp

Status

**Agent Delivery Events** 

| Intermediary Delivery Events | Status | Timestamp |
|---|---|---|
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent | Hashed/Encrypted | 3/16/2022 12:21:16 PM |
| Certified Delivered | Security Checked | 3/16/2022 12:23:00 PM |
| Signing Complete | Security Checked | 3/16/2022 12:23:56 PM |
| Completed | Security Checked | 9/23/2022 3:45:26 PM |
| Payment Events | Status | Timestamps |
| · | Otatus | · |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Rho, Inc. (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

### Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

| How to contact |
|---|
| may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows: To contact us by email send messages |
| To advise |
| To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address. |
| If you created a DocuSign account, you may update it with your new email address through your |

### To request paper copies from

account preferences.

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to an email to an email to an email to an email to an email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

## To withdraw your consent with

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to an and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

### Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

### Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send
  this Electronic Record and Disclosure to a location where you can print it, for future
  reference and access; and
- Until or unless you notify as a described above, you consent to receive exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you by during the course of your relationship with

# ACKNOWLEDGEMENT AND SIGNATURE SHEET

| Approved: |
|--------------------|
| Signature and Date |

| Approved: | Approved: |
|--------------------|--------------------|
| Signature and Date | Signature and Date |

| Approved: | Approved: |
|-----------------------|-----------------------|
| Judith James, MD, PhD | Meggan Mackay, MD, MS |
| Protocol Co-Chair | Protocol Co-Chair |
| Signature and Date | Signature and Date |


| Approved: | Approved: |
|--------------------------|------------------------|
| Dinesh Khanna, MBBS, MSC | Amit Bar-Or, MD, FRCPC |
| Protocol Co-Chair | Protocol Co-Chair |
| Signature and Date | Signature and Date |
| | March 16 2022 |

| Approved: | Approved: |
|----------------------|--------------------|
| Virginia Pascual, MD | Stacy Ardoin, MD |
| Protocol Co-Chair | Protocol Co-Chair |
| Signature and Date | Signature and Date |

| Approved: | Approved: |
|---------------------------|--------------------|
| Natasha Mckerran Ruth, MD | Tracey Wright, MD |
| Protocol Co-Chair | Protocol Co-Chair |
| Signature and Date | Signature and Date |